CLINICAL TRIAL: NCT01095536
Title: The Observational Cohort Study to Identify Risk Factors for Shoulder Pain and Emesis After Laparoscopic Cholecystectomy Under General Anesthesia
Brief Title: Risk Factors for Shoulder Pain and Emesis After Laparoscopic Cholecystectomy
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Taipei Veterans General Hospital, Taiwan (Other Government)
Responsible Party: Chiu-Ming Ho, M.D., Ph.D./Associate Professor and Attending Anesthesiologist, Department of Anesthesiology, Taipei Veterans General Hospital, Taipei, Taiwan
Other Study IDs: 201001019IC
Record Dates: First submitted 2010-03-28; First posted 2010-03-30 (Estimated); Last update posted 2010-10-06 (Estimated); Status verified 2010-03

CONDITIONS: Shoulder Pain; Nausea; Vomiting
Keywords: laparoscopic cholecystectomy, elective; anesthesia, general; shoulder pain; nausea; vomiting; laparoscopic cholecystectomy; general anesthesia
MeSH Terms: conditions — Shoulder Pain; Nausea; Vomiting

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Risk factors for postoperative shoulder pain after laparoscopic cholecystectomy were not clear. Moreover, risk factors for postoperative emesis specially for this surgery were not detailed and accurate. The present study is a prospective cohort study to identify risk factors for shoulder pain and emesis within 24 hours in Chinese patients after laparoscopic cholecystectomy under general anesthesia.

DETAILED DESCRIPTION:
The present study is a prospective cohort study to identify risk factors for shoulder pain and emesis within 24 hours in Chinese patients after laparoscopic cholecystectomy under general anesthesia.

ELIGIBILITY:
Inclusion Criteria:

* > 21 years old,
* Chinese patient

Exclusion Criteria:

* current pregnancy,
* patients with history of upper laparotomy,
* inability to communicate before operation,
* persistent emesis or shoulder pain before operation,
* patients who converted to open cholecystectomy,
* receiving postoperative ventilator support,
* unstable postoperative condition or major complications.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients scheduled for elective laparoscopic cholecystectomy
Sampling Method: Non-Probability Sample
Enrollment: 380 (Estimated)
Dates: Start 2010-02; Primary Completion 2011-02 (Estimated); Study Completion 2011-02 (Estimated)

PRIMARY OUTCOMES:
incidence of postoperative shoulder pain and emesis | within postoperative 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: Chiu-Ming Ho, M.D., Ph.D., Principal Investigator — Department of Anesthesiology, Taipei Veterans General Hospital, Taipei, Taiwan
Locations (1):
- Department of Anesthesiology, Taipei Veterans General Hospital, Taipei, Taiwan, Taiwan